CLINICAL TRIAL: NCT06383936
Title: FAldini Sport Total Joint Arthroplasty-Knee II: Toward Rehabilitation of Sports Activity Following Total Knee Arthroplasty
Brief Title: FAldini Sport Total Joint Arthroplasty-Knee II
Acronym: FAST-K II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST-K II
Record Dates: First submitted 2024-04-11; First posted 2024-04-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TKA patients (Experimental)
  Interventions: Procedure: intensive rehabilitation after uncemented TKA

INTERVENTIONS:
Procedure: intensive rehabilitation after uncemented TKA — patients undergoing an intensive rehabilitation protocol after uncemented tka

SUMMARY:
The majority of patients undergoing total knee arthroplasty are elderly individuals with low functional demands, aiming to alleviate pain. However, there exists a subgroup of younger patients, under the age of 65, with higher functional demands. The purpose of this study is to evaluate the return to sports activities in this patient group following a non-cemented total knee arthroplasty procedure and a specific rehabilitation protocol. The investigators expect that with the use of non-cemented prostheses and a specific rehabilitation protocol, many of these patients will safely resume sports activities.

DETAILED DESCRIPTION:
Most of the patients requiring total knee arthroplasty (TKA) suffer from primary geriatric osteoarthritis. These are predominantly elderly women, often overweight. According to the 2020 RIPO report, the average age of patients receiving primary bi- or tri-compartment knee replacement implants is 70.5 years, with 70% being women, 84% suffering from primary osteoarthritis; 40% are overweight, and 42% are obese. Generally, these individuals are frail elderly with almost complete immobility due to arthritis; post-surgery, relieved of pain, these patients typically return to very modest physical activity in terms of duration and intensity.

However, there exists a wholly different subgroup. These are patients aged ≤65 years, often men, who have been engaged in one or more sports activities since youth. Often, due to a sports-related injury, patients present to orthopedic consultation at a much younger age, with a severely arthritic condition, such as from ligamentous or meniscal trauma rendering the knee less stable, yet these patients have continued to load it intensely during sports activities. Literature and registry studies indicate that the incidence of TKA in this ≤65 age group has recently increased and is expected to rise further. Almost all of these patients have an ambitious postoperative recovery expectation, aiming to return to sports practice. This expectation is generally unmet today because the entire clinical pathway is typically designed for the first subgroup described above, the elderly and frail.

With the use of cemented knee prostheses, which remain the most commonly adopted choice worldwide, the overload on the implant leads to an increased incidence of aseptic loosening at the prosthesis-cement interface. This results in poor clinical and functional outcomes in the athletic patient subgroup and an increased failure rate, necessitating prosthetic revision, which is even more invasive and costly. Modern uncemented TKAs involve initial stable implant fixation through a robust press-fit mechanism of the component to bone and additional pegs for added stability. Definitive biological stability is achieved around 12 weeks post-surgery through osseointegration at the prosthesis interface facilitated by highly porous and/or hydroxyapatite-coated component surfaces.

Uncemented TKAs have shown undeniable advantages over the years, including reduced surgical time (with consequent reduction in general and infection-related complications), preservation of bone stock, and greater ease of performing prosthetic revision procedures. Additionally, with next-generation uncemented prostheses, the problem of loosening at the interface has significantly diminished, thanks to the use of biomaterials allowing firm implant fixation over time, enabling a quicker and more efficient patient activity resumption with a lower risk of prosthetic overload damage.

The long-term goal of this project is to explore whether and under what conditions it is possible to envision a return to sports activity for individuals who have undergone TKA. This type of intervention would constitute a form of tertiary prevention, aimed at containing and controlling the complex outcomes of a pathology, in this case, the drastic reduction in quality of life caused by the suspension of sports practice for this population subgroup. The larger the affected population, the more significant the importance of tertiary prevention, and thus the better the final outcome.

Regular physical activity is a well-known protective factor for the prevention and management of non-communicable diseases. According to the latest WHO (World Health Organization) guidelines from 2020, in adults (18-65 years), physical activity confers benefits for several health outcomes, reducing overall mortality, cardiovascular disease mortality, incidence of hypertension, breast and colon cancer, and type 2 diabetes onset. Physical activity also has mental health benefits, delays dementia onset, can contribute to maintaining a healthy weight, and overall well-being. It also helps prevent falls and fall-related injuries, as well as slowing down bone health decline and functional capacity decline.

The aim of our study is to evaluate the clinical and functional outcomes in patients aged 40 to 65 undergoing uncemented TKA with functional alignment and subjected to an intensive rehabilitation protocol aimed at returning to sports activity at the two orthopedic units, "Orthopedic and Traumatological Clinic 1" and "Orthopedics-Traumatology and Prosthetic Surgery and Hip and Knee Reimplantation"

ELIGIBILITY:
Inclusion Criteria:

* aged between 40 and 65 years,
* both men and women,
* individuals who engaged in sports until knee pathology hindered them. - "Saltin-Grimby Physical Activity Level Scale" 3 or 4.

Exclusion Criteria:

* Patients with rheumatic and/or neuromuscular disorders.
* Patients with extreme knee deformity.
* Patients with secondary osteoarthritis with compromised bone quality.
* Patients with coronal knee instability.
* Pregnant patients.
* Patients with medical conditions or physical conditions incompatible with the use of magnetic resonance imaging and electrostimulation (active and passive implanted biomedical devices, epilepsy, severe venous insufficiency in the lower limbs).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
number of patients returning to sports activities assessed by questionnaire | 1 year from the surgery
clinical and functional outcomes measured as the variation in the Knee Society Score | at 1, 3, 6 and 12 months from the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy